CLINICAL TRIAL: NCT02652416
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses and Multiple Oral Doses of BI 1026706 in Healthy Chinese and Japanese Male Volunteers (Randomised, Double-blind, Placebo-controlled Trial)
Brief Title: Safety, Tolerability and Pharmacokinetics of BI 1026706 in Healthy Chinese and Japanese Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1320.23
Record Dates: First submitted 2016-01-08; First posted 2016-01-11 (Estimated); Results first posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- SRD part (low dose) (Experimental): Chinese, Japanese both
  Interventions: Drug: BI 1026706
- SRD part (medium dose) (Experimental): Chinese, Japanese both
  Interventions: Drug: BI 1026706
- SRD part (high dose) (Experimental): Chinese, Japanese both
  Interventions: Drug: BI 1026706
- MD part (high dose) (Experimental): Chinese, Japanese both
  Interventions: Drug: BI 1026706
- Placebo (SRD part) (Experimental): placebo
  Interventions: Drug: Placebo
- Placebo (MD part) (Placebo Comparator): placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1026706 — oral administration
  Arms: MD part (high dose); SRD part (high dose); SRD part (low dose); SRD part (medium dose)
Drug: Placebo — placebo
  Arms: Placebo (MD part); Placebo (SRD part)

SUMMARY:
Safety and tolerability of BI 1026706 in healthy Chinese and Japanese male subjects following oral administration of single rising doses (SRD) followed by multiple rising doses (MRD)

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (BP, PR), 12-lead ECG, and clinical laboratory tests
* Chinese ethnicity or Japanese ethnicity, according to the following criteria:
* Chinese; born in China or ethnic Chinese born outside of China, and a descendent of 4 ethnic Chinese grandparents who were all born in China
* Japanese; born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who were all born in Japan
* Age of 20 to 45 years (incl.) - BMI of 18.5 to 25 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good clinical practice (GCP) and local legislation.- Male subjects who agree to minimize the risk of female partners becoming pregnant by fulfilling any of the following criteria starting from at least 30 days before the first administration of trial medication and until 30 days after trial completion:
* Use of adequate contraception, e.g. any of the following methods plus condom: combined oral contraceptives, intrauterine device
* Vasectomised (vasectomy at least 1 year prior to enrolment)
* Surgically sterilised (including hysterectomy) female partner

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) is deviating from normal and judged as clinically relevant by the investigator
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract that could interfere with kinetics of the trial medication (except appendectomy and simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections including HIV, viral hepatitis and (or) tuberculosis or evidence of tuberculosis infection as defined by a positive QuantiFERON TB-Gold (or T-SPOT) test. Subjects with a positive QuantiFERON TB-Gold (or T-SPOT) test may participate in the study if further work up (according to local practice/guidelines) establishes conclusively that the subject has no evidence of active tuberculosis. If presence of latent tuberculosis is established, then treatment must have been initiated and maintained according to local country guidelines.
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Intake of biologic agents other than current study medication or drugs considered likely to interfere with the safe conduct of the study
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial or that might prolong the QT/QTc interval
* Participation in another trial (including bioequivalence trial) with an investigational drug within 90 days or 5 half-lives (whichever is greater) prior to planned administration of trial medication
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 30 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 200 mL within 30 days prior to administration of trial medication or intended donation during the trial
* Intention to perform excessive physical activities within one week prior to administration of trial medication or during the trial
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms) or any other relevant ECG finding at screening
* A history of additional risk factors for Torsades de Pointes (such as heart failure, hypokalemia, or family history of Long QT Syndrome)
* Have received any live bacterial or live viral vaccination in the 12 weeks prior to the date of screening. Subjects must agree not to receive a live bacterial or live viral vaccination during the study and up to 12 months after the last administration of study drug
* Have received Bacille Calmette-Guerin (BCG) vaccination in the 12 months prior to the date of screening. Subjects must agree not to receive BCG vaccination during the study and up to 12 months after the last administration of study drug
* Male patients who do not agree to minimize the risk of female partners becoming pregnant from at least 30 days before the first administration of trial medication and until 30 days after trial completion.
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because considered not able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-09-16 (Actual); Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Souseikai Hakata Clinic, Fukuoka, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blind, placebo-controlled, single-centre trial investigating single rising dose (SRD) groups (25 milligram (mg), 50 mg and 100 mg) and a multiple dose (MD) (100 mg) in healthy Chinese and Japanese male subjects. This trial had an SRD plus MD nested design. All subjects from SRD 100 mg also participated in the MD part.
Pre-assignment Details: Only subjects that met all the study inclusion and none of the exclusion criteria were to be entered in the study. All subjects were free to withdraw from the clinical trial at any time for any reason given. Close monitoring of all subjects was adhered to throughout the trial conduct. Rescue therapies was allowed for all subjects as required.
Groups:
- Placebo: The subjects were administered film-coated tablets matching placebo orally with 240 milliliter (mL) water after an overnight fast of at least 10 hours (h).
- BI 1026706 25 mg: The subjects were administered 25 mg film-coated tablet single dose orally with 240 mL water after an overnight fast of at least 10h.
- BI 1026706 50 mg: The subjects were administered 50 mg [25 mg*2] film-coated tablets single dose orally with 240 mL water after an overnight fast of at least 10h.
- BI 1026706 100 mg: The subjects were administered 100 mg film-coated tablet [SRD] as single dose followed with 100 mg film-coated tablets [MD] twice daily for 11 days with a final single dose in the morning of Day 12 orally with 240 mL water after an overnight fast of at least 10h.
Period: Overall Study
Arm/Group | Placebo | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Started | 18 | 18 | 18 | 18
Subjects Who Participated in MD Part (All subjects who participated in the 100 mg dose group of SRD part continued in the MD part) | 6 | 0 | 0 | 18
Completed | 18 | 18 | 18 | 18
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS) : This subject set included all subjects who were dispensed study medication and were documented to have taken at least 1 dose of investigational treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg | Total
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 72
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.4 (7.74) | 28.6 (7.83) | 26.4 (5.72) | 28.1 (5.40) | 28.4 (6.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 18 | 18 | 18 | 18 | 72

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Drug-related Adverse Events (AEs)
Description: The percentage of subjects with drug-related AEs indicate the safety and tolerability of BI 1026706 in healthy Chinese and Japanese male subjects following oral administration of single rising doses of 25 mg, 50 mg, and 100 mg, followed by multiple doses of 100 mg bid.
Time Frame: From first drug administration to 4 days after last drug intake, up to 19 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Number analyzed (Participants) | 18 | 18 | 18 | 18
Percentage of participants | 0.0 | 0.0 | 0.0 | 5.6

2. Secondary Outcome: Cmax
Description: This outcome measure presents maximum measured concentration of the analyte [BI 1026706] in plasma.
  TS-SRD part: This subject set included all subjects who were dispensed BI 1026706 and were documented to have taken at least 1 dose of investigational treatment in the SRD part. All subjects in the TS-SRD part who provided at least 1 PK parameter in the SRD part that was not excluded were to be considered for this endpoint.
Time Frame: -1:30 (hours:minutes) before drug administration and 0:15, 0:30, 0:45, 1:00, 1:30, 2:00, 2:30, 3:00, 4:00, 6:00, 8:00, 10:00, 12:00, 24:00, 34:00, 48:00 and 72:00 (hours:minutes) after drug administration.
Population: PharmacoKinetic Set (PKS)-SRD part: This set included all evaluable subjects of the TS-SRD part who were administered BI 1026706, and provided at least 1 observation for at least 1 pharmacokinetic (PK) secondary endpoint without important protocol violations relevant for the evaluation of PK secondary endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nmol)/Liter (L)
Groups:
- BI 1026706 100 mg: The subjects were administered 100 mg film-coated tablet single dose orally with 240 mL water after an overnight fast of at least 10h.
Arm/Group | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Number analyzed (Participants) | 18 | 18 | 18
nanomole (nmol)/Liter (L)
  Chinese: number analyzed (Participants) | 9 | 9 | 9
  Chinese | 298 (42.8) | 677 (54.6) | 1120 (45.7)
  Japanese: number analyzed (Participants) | 9 | 9 | 9
  Japanese | 338 (45.5) | 595 (30.3) | 900 (51.2)

3. Secondary Outcome: Tmax
Description: This outcome measure presents time from dosing to maximum measured concentration of the analyte [BI 1026706] in plasma.
  All subjects in the TS-SRD part who provided at least 1 PK parameter in the SRD part that was not excluded were to be considered for this endpoint.
Time Frame: as for outcome 2
Population: PKS-SRD part.
Measure: Median (Full Range); unit: h
Arm/Group | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Number analyzed (Participants) | 18 | 18 | 18
h
  Chinese: number analyzed (Participants) | 9 | 9 | 9
  Chinese | 2.50 [0.75 to 4.00] | 1.50 [1.00 to 2.00] | 2.00 [0.75 to 4.00]
  Japanese: number analyzed (Participants) | 9 | 9 | 9
  Japanese | 3.00 [1.00 to 4.00] | 4.00 [0.75 to 4.00] | 3.00 [1.00 to 4.00]

4. Secondary Outcome: AUC0-12
Description: This outcome measure presents area under the concentration-time curve of the analyte [BI 1026706] in plasma over the time interval from 0 extrapolated to 12 hours (AUC0-12).
  All subjects in the TS-SRD part who provided at least 1 PK parameter in the SRD part that was not excluded were to be considered for this endpoint.
Time Frame: as for outcome 2
Population: PKS-SRD part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Number analyzed (Participants) | 18 | 18 | 18
nmol*h/L
  Chinese: number analyzed (Participants) | 9 | 9 | 9
  Chinese | 1340 (51.0) | 3260 (62.1) | 5340 (42.4)
  Japanese: number analyzed (Participants) | 9 | 9 | 9
  Japanese | 1650 (43.5) | 3270 (31.5) | 4620 (45.4)

5. Secondary Outcome: AUC0-infinity
Description: This outcome measure presents area under the concentration-time curve of the analyte [BI 1026706] in plasma over the time interval from 0 extrapolated to infinity.
  All subjects in the TS-SRD part who provided at least 1 PK parameter in the SRD part that was not excluded were to be considered for this endpoint.
Time Frame: as for outcome 2
Population: PKS-SRD part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Number analyzed (Participants) | 18 | 18 | 18
nmol*h/L
  Chinese: number analyzed (Participants) | 9 | 9 | 9
  Chinese | 1830 (45.9) | 4170 (59.1) | 7350 (37.1)
  Japanese: number analyzed (Participants) | 9 | 9 | 9
  Japanese | 2290 (40.4) | 4240 (29.7) | 6500 (37.7)

6. Secondary Outcome: t1/2
Description: This outcome measure presents terminal half-life of the analyte [BI 1026706] in plasma.
  All subjects in the TS-SRD part who provided at least 1 PK parameter in the SRD part that was not excluded were to be considered for this endpoint.
Time Frame: as for outcome 2
Population: PKS-SRD part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h
Arm/Group | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Number analyzed (Participants) | 18 | 18 | 18
h
  Chinese: number analyzed (Participants) | 9 | 9 | 9
  Chinese | 11.5 (70.3) | 9.44 (37.3) | 13.6 (64.6)
  Japanese: number analyzed (Participants) | 9 | 9 | 9
  Japanese | 14.3 (65.4) | 8.86 (56.4) | 12.3 (45.6)

7. Secondary Outcome: Cmax,ss
Description: This outcome measure presents maximum measured concentration of the analyte [BI 1026706] in plasma at steady state over a uniform dosing interval tau.
  TS-MD part: This subject set included all subjects from the 100 mg group in the SRD part who were dispensed BI 1026706 and were documented to have taken at least 1 dose of investigational treatment in the MD part. All subjects in the TS-MD part who provide at least 1 PK parameter in the MD part that was not excluded were to be considered for this endpoint.
Time Frame: 23:55, 47:55, 71:55, 95:55, 119:55, 167:55, 239:55, 263:55, 264:15, 264:30, 264:45, 265:00, 265:30, 266:00, 266:30, 267:00, 268:00, 270:00, 272:00, 274:00, 276:00, 288:00, 298:00, 312:00 and 336:00 (hours:minutes) after drug administration.
Population: PKS-MD part: This set included all evaluable subjects of the TS-MD part who were administered BI 1026706, and provided at least 1 observation for at least 1 PK secondary endpoint without important protocol violations relevant for the evaluation of PK secondary endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Groups:
- BI 1026706 100 mg: The subjects were administered 100 mg film-coated tablets twice daily for 11 days with a final single dose in the morning of Day 12 orally with 240 mL water after an overnight fast of at least 10h.
Arm/Group | BI 1026706 100 mg
Number analyzed (Participants) | 18
nmol/L
  Chinese: number analyzed (Participants) | 9
  Chinese | 1570 (36.5)
  Japanese: number analyzed (Participants) | 9
  Japanese | 1540 (25.7)

8. Secondary Outcome: Tmax,ss
Description: This outcome measure presents time from last dosing to maximum concentration of the analyte [BI 1026706] in plasma at steady state (tmax,ss) .
  All subjects in the TS-MD part who provide at least 1 PK parameter in the MD part that was not excluded were to be considered for this endpoint.
Time Frame: as for outcome 7
Population: PKS-MD part.
Measure: Median (Full Range); unit: h
Arm/Group | BI 1026706 100 mg
Number analyzed (Participants) | 18
h
  Chinese: number analyzed (Participants) | 9
  Chinese | 2.50 [0.750 to 3.00]
  Japanese: number analyzed (Participants) | 9
  Japanese | 2.00 [0.750 to 4.00]

9. Secondary Outcome: AUC Tau,ss
Description: This outcome measure presents area under the concentration-time curve of the analyte [BI 1026706] in plasma at steady state over a uniform dosing interval tau (AUC tau,ss).
  All subjects in the TS-MD part who provide at least 1 PK parameter in the MD part that was not excluded were to be considered for this endpoint.
Time Frame: as for outcome 7
Population: PKS-MD part.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | BI 1026706 100 mg
Number analyzed (Participants) | 18
nmol*h/L
  Chinese: number analyzed (Participants) | 9
  Chinese | 9390 (35.2)
  Japanese: number analyzed (Participants) | 9
  Japanese | 8550 (26.4)

ADVERSE EVENTS:
Time Frame: From first drug administration to 4 days after last drug intake, up to 19 days.
Description: This trial had an SRD plus MD nested design. All subjects from SRD 100 mg also participated in the MD part.
Arm/Group | Placebo | BI 1026706 25 mg | BI 1026706 50 mg | BI 1026706 100 mg
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18 | 2/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=18) | BI 1026706 25 mg (N=18) | BI 1026706 50 mg (N=18) | BI 1026706 100 mg (N=18)
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.